CLINICAL TRIAL: NCT04138966
Title: Nociceptive Monitoring With Skin Conductance and Nol-index in Moderate-to-high Risk Cardiovascular Patients
Brief Title: Comparing Skin Conductance and Nol-index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2019/427Am1
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Analgesia; Anesthesia; Monitoring; Vascular Diseases; Cardiac Disease
MeSH Terms: conditions — Agnosia; Vascular Diseases; Heart Diseases | interventions — Galvanic Skin Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing general anesthesia: Patients are monitored with Nol-Index, skin conductance, and antinociception-index
  Interventions: Device: Nol-Index; Device: Skin Conductance

INTERVENTIONS:
Device: Nol-Index — Multiparametric monitor that studies that establishes an index as a surrogate to nociception
  Other Names: PMD-200
Device: Skin Conductance — Measures skin conductance as a surrogate to nociception
  Other Names: The PainMonitor Index

SUMMARY:
Comparison of twà different nociception monitors during general anesthesia

DETAILED DESCRIPTION:
Analgesia remains a challenge in anesthesia. Several monitors have shown potential in detecting insufficient analgesia during general anesthesia, but they have not been investigated in patients undergoing cardiac and vascular surgery. In this study, we will compare skin conductance (Medstorm, Norway) and nol-index (Medasense, Israel) w during noxious and non-noxious stimuli. This study is carried out on patients included in another study (Nol-Index Guided Remifentanil Analgesia Versus Standard Analgesia During Moderate-to-High Risk Cardiovascular Surgery).

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-high risk cardiac or vascular surgery
* ASA 2-4

Exclusion Criteria:

* chronic arrhythmia (e.g. atrial fibrillation)
* aortic insufficiency
* pacemaker
* implanted defibrillator
* valve surgery

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac or vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Nol-Index response | 1 to 2 hours
  Nol-Index (diminsenliss value from 0 to 100) will be assessed during noxious and non noxious stimuli
Skin conductance response | 1 to 2 hours
  Peaks per second change during noxious and non noxious stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Luc Barvais, MD, PhD, Principal Investigator — Anesthesia Department, Erasme Hospital
Locations (1):
- Anesthesia Department, Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided